CLINICAL TRIAL: NCT04396678
Title: Developing a PrEP Adherence Intervention Targeting At-Risk and Substance Using Women
Acronym: PEARL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Baltimore City Health Department (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 126993
Record Dates: First submitted 2020-03-26; First posted 2020-05-20 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PrEP Standard of Care (No Intervention): PrEP standard of care, administered through the Baltimore City Health Department
- PrEP standard of care+behavioral intervention (Experimental): PrEP standard of care, administered through the Baltimore City Health Department, and the behavioral intervention.
  Interventions: Behavioral: PrEP standard of care+behavioral intervention

INTERVENTIONS:
Behavioral: PrEP standard of care+behavioral intervention — The intervention includes three main components: 1) group PrEP engagement sessions, which include four educational sessions that situate PrEP in a broader framework of access and barriers to care, provider/patient communication, sexual health, HIV/STI education, harm reduction around drug use, stigma, risk compensation and safe sex, and health/science literacy; 2) peer navigation, which aims to help women navigate healthcare engagement with the SPARC nurse practitioner and other providers; and 3) an mHealth component, consisting of a two-way text messaging system through which women will receive automated daily messages and weekly messages requesting adherence reports.
  Arms: PrEP standard of care+behavioral intervention

SUMMARY:
The purpose of this study is to develop and assess the feasibility, acceptability, and preliminary efficacy on adherence of a community-informed intervention for tenofovir/emtricitabine (TDF/FTC) pre-exposure prophylaxis (PrEP) engagement among street-based female sex workers (FSW) in Baltimore, Maryland.

DETAILED DESCRIPTION:
This study is a prospective two-group trial comparing the efficacy of a comprehensive PrEP adherence program compared to PrEP standard of care among FSW. Outcomes will be assessed through self-reported PrEP adherence as well as biological adherence indicators.

The intervention includes three main components: 1) group PrEP engagement sessions, which include four educational sessions that situate PrEP in a broader framework of access and barriers to care, provider/patient communication, sexual health, HIV/sexually transmitted infection (STI) education, harm reduction around drug use, stigma, risk compensation and safe sex, and health/science literacy; 2) peer navigation, which aims to help women navigate healthcare engagement with the SPARC nurse practitioner and other providers; and 3) an mHealth component, consisting of a two-way text messaging system through which women will receive automated daily messages and weekly messages requesting adherence reports.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Assigned female at birth and identify as a woman
* Traded sex for money or drugs at least three times in the past three months
* HIV negative
* Willing to initiate PrEP
* Not knowingly pregnant or planning to become pregnant during the following 6 months.

Exclusion Criteria:

* Currently taking PrEP for HIV prevention
* Inability to provide informed consent in English
* Women who are determined as too high or drunk
* Women who are cognitively impaired
* Does not agree to data sharing with the Baltimore City Health Department

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Currently identify as a woman or female
Enrollment: 39 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change over time to adherence to PrEP using plasma | 3 and 6 months
  Adherence as the biological outcome, measured by the use of plasma to see concentration of tenofovir (ng/mL), to examine the pilot study's impact on adherence and inform metrics and outcomes of a future R01.
Change over time to adherence to PrEP using dried blood spots | 3 and 6 months
  Adherence as the biological outcome, measured by the use of dried blood spots to see concentration of tenofovir (fmol/punch), to examine the pilot study's impact on adherence and inform metrics and outcomes of a future R01.

SECONDARY OUTCOMES:
Behavioral outcomes change over time | 3 and 6 months
  unsafe syringe use, unsafe sex, measured by survey. No scales for these, just individual questions about behavior. Syringe use are binary yes/no questions, condom use is frequency of condom use during vaginal, oral, and anal sex (separately).
Social outcomes change over time | 3 and 6 months
  Social support, measured by survey. Social support: Moser, A., Stuck, A. E., Silliman, R. A., Ganz, P. A., & Clough-Gorr, K. M. (2012). The eight-item modified Medical Outcomes Study Social Support Survey: psychometric evaluation showed excellent performance. Journal of clinical epidemiology, 65(10), 1107-1116.
  Possible range is 0-32, higher score indicates better outcome
Structural vulnerabilities change over time | 3 and 6 months
  housing, access to healthcare, measured by survey. Access to healthcare partially measured by: modified Kalichman, S. C., Catz, S., and Ramachandran, B. (1999). Barriers to HIV/AIDS treatment and adherence among African-American adults with disadvantaged education. Journal of the National Medical Association, 91, 439-446.
  Higher # endorsed means greater barriers to care
Individual health change over time | 3 and 6 months
  PrEP uptake, awareness and knowledge, measured by survey. Adapted from the ACTG Adherence Questionnaire The AIDS Clinical Trials Group (ACTG) (2009). ACTG Adherence Questionnaires. Retrieved at: https://prevention.ucsf.edu/sites/prevention.ucsf.edu/files/uploads/tools/surveys/pdf/2098.4188.pdf
  Independently developed self-report questions to measure PrEP uptake, knowledge, and perceived barriers and facilitators
Individual PrEP change over time | weekly, from baseline visit to last study visit (six months from baseline)
  PrEP adherence, measured by mHealth. Survey question: How many times in the past week have you taken your medication? Please respond with 0-7.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sherman, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- SPARC Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share data outside of the research plan